CLINICAL TRIAL: NCT00559845
Title: Phase II, Open Label, Neoadjuvant Study of Bevacizumab in Patients With Inflammatory or Locally Advanced Breast Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Patients With Inflammatory or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19884; 2006-003291-35 (EudraCT Number)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Epirubicin; Cyclophosphamide; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): Participants will receive FEC, followed by paclitaxel, given concomitantly with bevacizumab for approximately 3-12 months.
  Interventions: Drug: 5-fluorouracil; Drug: Epidoxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Biological: Bevacizumab

INTERVENTIONS:
Drug: 5-fluorouracil — 600 milligrams per meter squared (mg/m^2) as an intravenous (i.v.) bolus over ≤15 minutes every 3 weeks for 4 cycles.
Drug: Epidoxorubicin — 90 mg/m^2 as an i.v. infusion over 1 hour every 3 weeks for 4 cycles.
Drug: Cyclophosphamide — 600 mg/m^2 as an i.v. infusion over 1 hour every 3 weeks for 4 cycles.
Drug: Paclitaxel — Paclitaxel was administered at 80 mg/m^2 i.v. over 1 hour weekly for 12 weeks.
Biological: Bevacizumab — Bevacizumab was administered at 10 milligrams per kilogram (mg/kg) i.v. every 2 weeks for 6 cycles.
  Other Names: Avastin®

SUMMARY:
This single arm study will assess the efficacy and safety of sequential neoadjuvant chemotherapy and bevacizumab (Avastin), before surgery and/or radiotherapy, in participants with inflammatory or locally advanced operable breast cancer. Participants will receive 5-fluorouracil, epidoxorubicin and cyclophosphamide (FEC), followed by paclitaxel, given concomitantly with bevacizumab. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female participants, >=18 years of age;
* stage III, or inflammatory breast cancer;
* estrogen receptor/progesterone receptor (ER/PgR) positive or negative and human epidermal growth factor receptor 2 (HER-2) negative;
* normal left ventricular ejection fraction (LVEF).

Exclusion Criteria:

* previous chemotherapy/endocrine therapy;
* evidence of distant metastatic disease;
* other primary tumors in last 5 years (except for adequately treated cancer in situ of the cervix, or basal cell skin cancer);
* chronic daily treatment with >325 milligram per day (mg/day) aspirin, or >75mg/day clopidogrel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Italy (8):
  - Napoli, Campania
  - Reggio Emilia, Emilia-Romagna
  - Pordenone, Friuli Venezia Giulia
  - Genoa, Liguria
  - Mantova, Lombardy
  - Cuneo, Piedmont
  - Turin, Piedmont
  - Negrar, Veneto

REFERENCES:
- [Derived] Clavarezza M, Turazza M, Aitini E, Saracchini S, Garrone O, Durando A, De Placido S, Bisagni G, Levaggi A, Bighin C, Restuccia E, Scalamogna R, Galli A, Del Mastro L. Phase II open-label study of bevacizumab combined with neoadjuvant anthracycline and taxane therapy for locally advanced breast cancer. Breast. 2013 Aug;22(4):470-5. doi: 10.1016/j.breast.2013.03.012. Epub 2013 May 1. PMID 23642526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 participants were enrolled in 8 centers in Italy.
Groups:
- Bevacizumab: 5-fluorouracil, epidoxorubicin and cyclophosphamide (FEC), followed by paclitaxel, given concomitantly with bevacizumab for approximately 3-12 months.
  FEC: 5-Fluorouracil 600 milligrams per meter squared (mg/m^2) intravenous (i.v.) bolus over ≤15 minutes (min); epirubicin 90 mg/m^2 i.v. infusion over 1 hour; cyclophosphamide 600 mg/m^2 i.v. infusion over 1 hour every 3 weeks for 4 cycles.
  Paclitaxel: 80 mg/m^2 i.v. over 1 hour weekly for 12 weeks.
  Bevacizumab: 10 milligrams per kilogram (mg/kg) i.v. every 2 weeks for 6 cycles.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 56
Completed | 49
Not Completed | 7
Not completed — Withdrew Consent | 1
Not completed — Disease Progression | 1
Not completed — Adverse Event | 3
Not completed — Did Not Attend Cycle 6 Hospital Visit | 1
Not completed — Premature Surgery-Investigator Decision | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) population, defined as all participants that were included in the trial and underwent surgery.
Groups:
- Bevacizumab: FEC, followed by paclitaxel, given concomitantly with bevacizumab for approximately 3-12 months.
  FEC: 5-Fluorouracil 600 mg/m^2 i.v. bolus over ≤15 min; epirubicin 90 mg/m^2 i.v. infusion over 1 hour; cyclophosphamide 600 mg/m^2 i.v. infusion over 1 hour every 3 weeks for 4 cycles.
  Paclitaxel: 80 mg/m^2 i.v. over 1 hour weekly for 12 weeks.
  Bevacizumab: 10 mg/kg i.v. every 2 weeks for 6 cycles.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.00 (9.279)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response Following Principle Investigator Review
Description: Pathological complete response was defined as absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy.
Time Frame: Up to 7.5 years
Population: Intention-to-Treat (ITT) population, defined as all participants that were included in the trial and underwent surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 56
percentage of participants | 23.2

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with a Complete Response (CR) or Partial Response (PR) as defined by the Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as the disappearance of all target lesions; PR was defined as a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Up to 7.5 years
Population: ITT population, defined as all participants that were included in the trial and underwent surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 56
percentage of participants | 59.0

3. Secondary Outcome: Percentage of Participants With Breast-Conserving Surgery
Description: Rate of breast conversing surgery is defined as percentage of participants who achieved breast conversing surgery out of the ITT population without inflammatory breast cancer, as these participants received mastectomy irrespective of their response to neoadjuvant treatment.
Time Frame: Up to 7.5 years
Population: ITT population, defined as all participants that were included in the trial and underwent surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 56
percentage of participants
  Breast-conserving | 17.0
  Breast-conserving Plus Axillary Dissection | 13.2

4. Secondary Outcome: Percentage of Participants With Disease-Free Interval
Description: Disease-free interval was defined as the time from enrollment until recurrence of tumor or death from any cause, and was estimated using the Kaplan-Meier method. The percentage of participants without events at Months 12, 24, 36, 48, and 60 is presented.
Time Frame: Months 12, 24, 36, 48, and 60
Population: ITT population, defined as all participants that were included in the trial and underwent surgery. Here, number of participants analyzed signifies those participants who were evaluable for the outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 53
percentage of participants
  12 Months | 92.2 [85.1 to 99.8]
  24 Months | 84.3 [74.9 to 94.9]
  36 Months | 80.4 [70.2 to 92.1]
  48 Months | 76.5 [65.7 to 89.1]
  60 Months | 76.5 [65.7 to 89.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from enrollment of participant to death from any cause.
Time Frame: Up to 7.5 years
Population: Data for the outcome measure was not collected.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Experiencing Any Adverse Event
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 7.5 years
Population: Safety population, defined as all participants who received at least one infusion of Bevacizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 56
percentage of participants | 100.0

ADVERSE EVENTS:
Time Frame: Up to 7.5 years
Description: Safety population defined as all participants who received at least one infusion of Bevacizumab.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 8/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=54)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Retinopathy Hypertensive (Eye disorders) | 1
Febrile Infection (Infections and infestations) | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1
Cardiac Imaging Procedure Abnormal (Investigations) | 1
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Suicide Attempt (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=54)
Neutropenia (Blood and lymphatic system disorders) | 22
Leukopenia (Blood and lymphatic system disorders) | 15
Anaemia (Blood and lymphatic system disorders) | 12
Conjunctivitis (Eye disorders) | 9
Nausea (Gastrointestinal disorders) | 38
Diarrhea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 11
Abdominal Pain Upper (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 6
Haemorrhoids (Gastrointestinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 30
Mucosal Inflammation (General disorders) | 18
Pyrexia (General disorders) | 15
Oedema (General disorders) | 3
Pain (General disorders) | 3
Alanine Aminotransferase Increased (Investigations) | 6
Ast Increased (Investigations) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Bone Pain (Musculoskeletal and connective tissue disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Paraesthesia (Nervous system disorders) | 27
Headache (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 36
Nail Disorder (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 3
Astringent Therapy (Surgical and medical procedures) | 3
Hypertension (Vascular disorders) | 13
Phlebitis (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.